CLINICAL TRIAL: NCT06561737
Title: Effect of Video-Based Teaching on Urinary Catheterization Skills: Randomized Controlled Study
Brief Title: Effect of Video-Based Teaching on Urinary Catheterization Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hanife DURGUN, Assos. Prof. (Head of the Fundamentals of Nursing Department), Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Video effect
Record Dates: First submitted 2024-08-12; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Nursing Caries
Keywords: Nursing Caries; Urinary Chather; Nursing Students; Video
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: This study was a randomized, single-blind, parallel group-controlled trial.
Who Masked: Participant
Masking Description: The study was single-blind and the participants were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video group (Experimental): For the students in the experimental group, the application was first demonstrated on a model by the course instructor, after which each student was required to perform the application individually. While the students were performing the application, someone not part of the research team recorded them on their phones. During the application, two researchers independently assessed the student's skills using the application checklist. Afterward, the students were asked to watch their videos and evaluate themselves over a 15-day period. After 15 days, the students were called back and asked to perform the same application again. At this stage, the researchers once again evaluated the students independently.
  Interventions: Other: Video
- Control group (No Intervention): The process of insertion and removal of urinary catheterization was first explained to the students in the control group by the instructor of the course in the research team by demonstrations on the models. Then, each student was allowed to perform the application. Then, all students were invited again 15 days later for the second application. In both applications, the students were evaluated independently by the researchers.

INTERVENTIONS:
Other: Video — For the students in the experimental group, the application was first demonstrated on a model by the course instructor, after which each student was required to perform the application individually. While the students were performing the application, someone not part of the research team recorded them on their phones. During the application, two researchers independently assessed the student's skills using the application checklist. Afterward, the students were asked to watch their videos and evaluate themselves over a 15-day period. After 15 days, the students were called back and asked to perform the same application again. At this stage, the researchers once again evaluated the students independently.
  Arms: Video group

SUMMARY:
Urinary catheters, which can be urethral or suprapubic, are frequently used to measure urine output, control urinary output during surgery, and provide urine output in individuals with urinary excretion problems such as urinary incontinence and urinary retention (Chadha et al., 2024; Feneley, Hopley, & Wells, 2015). This practice, which has an important place in patient safety, should be explained to nursing students in line with current evidence-based knowledge, and students should have access to up-to-date information and improve their skills in this regard (Aldridge & Hummel, 2019; Güven Özdemir & Kaya, 2023). However, nursing students may not have the opportunity to perform this practice in the clinical field due to the high risk of infection and the fact that the practice requires more sensitivity in terms of privacy than many other practices (Aksoy & Paslı Gürdoğan, 2022; Chang, 2022; Güven Özdemir & Kaya, 2023). This situation may prevent students from reinforcing their knowledge and skills, and therefore, after graduation, newly graduated nurses may not have the opportunity to practice this practice in their working life (Aksoy & Paslı Gürdoğan, 2022; Chang, 2022; Güven Özdemir & Kaya, 2023).

DETAILED DESCRIPTION:
In nursing education, the combination of cognitive, psychomotor and attitudinal behaviors has an important place in the acquisition of professional skills. In the acquisition of psychomotor skills, educational teaching methods such as role playing, skill lists, simulator technologies, scenario-based trainings and video demonstrations are used (Filiz & Dikmen, 2017;McEnroe et al., 2020; Pivac et al., 2021). Smartphones and the internet, which have entered our lives with the developing technology, have led students to acquire new learning environments (McEnroe et al., 2020). Students have the opportunity to easily access the applications of the courses they want to research or watch on the internet. This situation has revealed the need to change the approach of today's nursing students to learning methods. Especially videos with skill-based trainings facilitate nursing students to learn skills (Mete & Uysal, 2010). The use of video demonstrations in education and training can make learning more enjoyable by visualizing the information as well as contributing to the reinforcement of the information learned, keeping it in memory and remembering it in the future. Using the video of the skill to be acquired in the learning process allows students to visualize and interpret the skill in their minds (Korhan et al., 2016).

Based on Bandura's Social Learning Theory and adapted from Applied Behavior Analysis, the Video Modeling Method aims for the individual to learn by observing. Video self-modeling practices are used for the acquisition of new skills, fluency in previously acquired skills, and reduction of problem behaviors. This practice first emerged in the early 1970s and its use in educational settings has been developing more slowly compared to other methods (Buggey & Ogle, 2012). This is a practice based on showing images of individuals performing the target behavior appropriately in order to enable them to exhibit new behaviors or skills (Dowrick & Hood, 1981).

It is very important for nursing students to recognize their own abilities, develop their skills and take responsibility for their learning. In a study investigating the methods preferred by undergraduate nursing students in learning the psychomotor skills required for clinical practice, students reported that clinical skills laboratory practice helped them learn on their own, they felt more sense of control and felt more confident in patient care (Ekeri Açıkgöz & Karaca, 2014).

As much as the learning methods used in education and training of nursing students, the evaluation of the developed skill, the student's ability to see the student's mistakes and to recognize these mistakes are as important as the learning methods used in education and training.

ELIGIBILITY:
Inclusion Criteria:

* A first-year student in the department of nursing,
* smartphone users,
* taking the nursing principles course for the first time, t
* those who volunteered to participate in the study.

Exclusion Criteria:

* Graduating from health vocational high school,
* having previous knowledge of urinary catheter placement skills,
* wanting to withdraw from the study at any stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Urinary System Information Test Score | Through study completion, an average of 2 months
  The questionnaire was prepared by the researcher based on the literature (Potter et al., 2022; Akın, 2021). The knowledge test consists of 20 multiple-choice questions about the urinary system (3 questions) and urinary system practices (17 questions). The lowest score to be obtained from the test is 0 and the highest score is 20. Before the test was applied to the students, expert opinion was obtained from five lecturers who are experts in the field of Nursing Principles. The test was finalized in line with the recommendations of the experts.

SECONDARY OUTCOMES:
Urinary Catheterization Insertion Skill Checklist Score | through study completion, an average of 2 months
  The form was created by the researchers in line with the literature to examine and evaluate students' urinary catheterization placement skills (Gündoğdu & Dikmen, 2020; Potter et al., 2020; Stein & Hollen, 2023; Ertuğrul, 2023). For the skill list consisting of 47 items in total, expert opinions were obtained from five expert faculty members in the field of Fundamentals of Nursing and two clinical nurses. According to the created guideline; 2 points were given to the response of "Correctly performed application", 1 point to the response of "Application whose order was confused" and 0 points to the response of "Forgotten application or application that was not performed correctly". The skill checklist used to evaluate the skill performance of the students included 3 steps related to pre-application preparation, 29 steps related to the application phase and 15 steps related to catheter removal. Students can get a minimum score of 0 and a maximum score of 94 points from the checklist.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanife Durgun, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Assured that the information will not be shared with anyone

REFERENCES:
- [Result] Aksoy B, Pasli Gurdogan E. Examining effects of the flipped classroom approach on motivation, learning strategies, urinary system knowledge, and urinary catheterization skills of first-year nursing students. Jpn J Nurs Sci. 2022 Apr;19(2):e12469. doi: 10.1111/jjns.12469. Epub 2022 Jan 4. PMID 34984830
- [Result] Aldridge MD, Hummel F. Nursing Students' Perceptions of Skills Learning: A Phenomenological Study. Nurse Educ. 2019 May/Jun;44(3):170-174. doi: 10.1097/NNE.0000000000000569. PMID 30028766
- [Result] Chadha J, Thakur N, Chhibber S, Harjai K. A comprehensive status update on modification of foley catheter to combat catheter-associated urinary tract infections and microbial biofilms. Crit Rev Microbiol. 2024 Mar;50(2):168-195. doi: 10.1080/1040841X.2023.2167593. Epub 2023 Jan 18. PMID 36651058
- [Result] Chang CL. Effect of Immersive Virtual Reality on Post-Baccalaureate Nursing Students' In-Dwelling Urinary Catheter Skill and Learning Satisfaction. Healthcare (Basel). 2022 Aug 5;10(8):1473. doi: 10.3390/healthcare10081473. PMID 36011130
- [Result] Feneley RC, Hopley IB, Wells PN. Urinary catheters: history, current status, adverse events and research agenda. J Med Eng Technol. 2015;39(8):459-70. doi: 10.3109/03091902.2015.1085600. Epub 2015 Sep 18. PMID 26383168
- [Result] Ozdemir NG, Kaya H. The effectiveness of high-fidelity simulation methods to gain Foley catheterization knowledge, skills, satisfaction and self-confidence among novice nursing students: A randomized controlled trial. Nurse Educ Today. 2023 Nov;130:105952. doi: 10.1016/j.nedt.2023.105952. Epub 2023 Aug 23. PMID 37639878
- [Result] Pivac S, Skela-Savic B, Jovic D, Avdic M, Kalender-Smajlovic S. Implementation of active learning methods by nurse educators in undergraduate nursing students' programs - a group interview. BMC Nurs. 2021 Sep 18;20(1):173. doi: 10.1186/s12912-021-00688-y. PMID 34535119